CLINICAL TRIAL: NCT04023682
Title: Proposal to Conduct a Study Assessing Whether ProvodineTM Decreases Contamination of Anesthesia Providers' Hands During General Anesthesia Procedures
Brief Title: ProvodineTM Decreases Hand Contamination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sundara Reddy (Other)
Collaborators: Microdermis Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sundara Reddy, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201312709
Record Dates: First submitted 2019-06-12; First posted 2019-07-17 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Hand Hygiene
Keywords: Hand hygiene; Provodine; Hand contamination

STUDY DESIGN:
Intervention Model Description: Anesthesia providers will serve as their own controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anesthesia Provider hands (Other): Each provider will serve as their own control.
  Control phase is at baseline using standard hygiene practices.
  Intervention phase will include the addition of Provodine hand sanitizer
  Interventions: Drug: Provodine Hand Sanitizer

INTERVENTIONS:
Drug: Provodine Hand Sanitizer — Intervention with Provodine
  Other Names: Provodine

SUMMARY:
The purpose of this study is to see whether Provodine, an FDA approved product, provides long-lasting protection on the hands of staff who provide anesthesia for patients. If this product does provide long-lasting protection, it could be used for hand hygiene in the operating room and it could help prevent infections after operations. Fifteen anesthesia providers (15 main operating room [MOR] and 5 ambulatory surgery center [ASC]) who agree to participate will participate in the pre-intervention and intervention periods. During the pre-intervention or baseline period, the investigators will do bag broth cultures of anesthesia providers' hands just before the start of their first case of the day . The participants will then rinse and dry their hands to remove the culture medium. The investigators will also obtain cultures after the first case of the day, and after the second case. During the intervention period (ProvodineTM; usual hand hygiene practice), the investigators obtain hand cultures from the same anesthesia providers at the beginning of the day. The participants will then then do a hand scrub with ProvodineTM. The investigators will obtain a second hand culture at this point and participants will rinse and dry their hands to remove the culture medium and then apply a small amount of ProvodineTM as a hand rub. The investigators will obtain cultures after the first case of the day, and after the second case of the day. If participants are still providing anesthesia to their second case 6 hours after they applied ProvodineTM, the participants will apply a small of ProvodineTM amount as a hand rub at this time.

For anesthesia providers in the ASC, the investigators will use the same protocol with the following exception. Because cases are likely to be shorter, the investigators will obtain the final cultures after the last case of the day or after the case that ends closest to 6 hours after ProvodineTM was applied in the morning.

DETAILED DESCRIPTION:
During the pre-intervention or baseline period, the investigators will do bag broth cultures of anesthesia providers' hands just before the start of their first case of the day (n =25). The participants will then rinse and dry their hands to remove the culture medium. The investigators will also obtain cultures after the first case of the day (n = 25), and after the second case (n = 25). During the intervention period (ProvodineTM; usual hand hygiene practice), the investigators obtain hand cultures from the same anesthesia providers at the beginning of the day (n =25). The participants will then then do a hand scrub with ProvodineTM. The investigators will obtain a second hand culture at this point and participants will rinse and dry their hands to remove the culture medium and then apply a small amount of ProvodineTM as a hand rub (n =25). The investigators will obtain cultures after the first case of the day (n = 25), and after the second case of the day (n = 25). If participants are still providing anesthesia to their second case 6 hours after they applied ProvodineTM, the participants will apply a small of ProvodineTM amount as a hand rub at this time. For anesthesia providers in the ASC, the investigators will use the same protocol with the following exception. Because cases are likely to be shorter, the investigators will obtain the final cultures after the last case of the day or after the case that ends closest to 6 hours after ProvodineTM was applied in the morning.

The study procedures will occur on two different work days for the participants: one for the control day and one for the intervention day. The study procedures will be done by the end of these two working days. There is no long-term followup.

ELIGIBILITY:
Inclusion Criteria:

- Must be an anesthesia provider at The University of Iowa Hospitals and Clinics

Exclusion Criteria:

- Are not an anesthesia provider at The University of Iowa Hospitals and Clinics

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Durgempudi Tripura, MD, Principal Investigator — University of Iowa; Loreen Herwaldt, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Anesthesia Provider Hands: Anesthesia Providers hands cultures with standard hand hygiene
  Provodine Hand Sanitizer: Intervention with Provodine
Period: Overall Study
Arm/Group | Anesthesia Provider Hands
Started | 31
Completed | 25
Not Completed | 6
Not completed — Clinical schedules did not allow continued participation | 6

BASELINE CHARACTERISTICS:
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Control Period-Count the Number of Baseline Colony Forming Units Cultured From Anesthesiologist's Hands
Description: Each subject of the study will serve as their own controls and a comparison will be made between the control phase of the study and the intervention phase of the study.
  Control portion of the study-usual hand hygiene practice but prior to the anesthesiologist's first case of the day, bag broth cultures will be obtained and the number of CFU's will be counted (T1).
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Groups:
- Anesthesia Provider Hands: Anesthesia Providers hands cultures with standard hand hygiene
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 31
Colony forming units | 589.3 (823.7)

2. Primary Outcome: Intervention Period-Count the Number of Baseline Colony Forming Units Cultured From Anesthesiologist's Hands
Description: During the intervention period, a bag broth culture was performed immediately after the anesthesiologist enter the operating suite. Provodine was applied to the participant's hands, rubbed into his/her skin, washed hands, and dried with a sterile towel. After this a second bag broth culture was obtained.
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Groups:
- Anesthesia Provider Hands: Anesthesia Providers hands cultures after use with Provodine hand sanitizer.
  Provodine Hand Sanitizer: Intervention with Provodine
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 25
Colony forming units | 788.9 (1051.3)

3. Secondary Outcome: Control Phase-Count and Compare the Number of CFU's After the First Case of the Day.
Description: After the first surgical case for the day, a bag broth culture was collected (T2) during the control phase from each individual anesthesia provider.
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 31
Colony forming units | 825.2 (1299.2)

4. Secondary Outcome: Interventional Phase-Count and Compare the Number of CFU's After the First Case of the Day.
Description: After the first surgical case for the day, a bag broth culture was collected (T2) during the interventional phase from each individual anesthesia provider.
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Groups:
- Anesthesia Provider Hands: Anesthesia Providers hands cultures after use with Provodine hand sanitizer.
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 25
Colony forming units | 248.9 (709.0)

5. Secondary Outcome: Control Phase-Count and Compare the Number of CFU's After the Second Case of the Day.
Description: After the second surgical case for the day, a bag broth culture was collected (T3) during the control phase from each individual anesthesia provider.
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 31
Colony forming units | 971.2 (1998.3)

6. Secondary Outcome: Interventional Phase-Count and Compare the Number of CFU's After the Second Case of the Day.
Description: After the second surgical case for the day, a bag broth culture was collected (T3) during the interventional phase from each individual anesthesia provider.
Time Frame: Average of 1 day
Measure: Mean (Standard Deviation); unit: Colony forming units
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 25
Colony forming units | 382.2 (793.4)

7. Secondary Outcome: Number of Providers/Participants Who Acquired a Pathogen or Commensal During the Day.
Description: Participants participated in both the control as well as the interventional phase of this study. The number of unique providers who acquired a pathogen during the course of their day are counted and reported.
Time Frame: Average of 1 day
Measure: Number; unit: participants
Groups:
- Anesthesia Provider Hands: Anesthesia Providers hands cultures
Arm/Group | Anesthesia Provider Hands
Number analyzed (Participants) | 31
participants
  Total Number-Unique participants | 11
  Pathogens-Control phase | 2
  Pathogens-Interventional phase | 3
  Commensals-Control phase | 3
  Commensals-Interventional phase | 3

ADVERSE EVENTS:
Arm/Group | Anesthesia Provider Hands
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

LIMITATIONS AND CAVEATS:
The number of days that elapsed between the control phase and the interventional phase from each individual provider who completed both phases ranged from 1 day to 83 days. In the control phase, 31 providers participated (20 male, 11 female). Six providers withdrew and did not complete the interventional phase (3 male, 3 female).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes